CLINICAL TRIAL: NCT02460003
Title: Effectiveness of Physiotherapy Program in Patients With Cluster Headache
Brief Title: Physiotherapy Program for Cluster Headache
Acronym: PhyCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: AG Clinic (Other)
Collaborators: Instituto de Investigación Hospital Universitario La Paz (Other); Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CH-Physiotherapy
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Physical Therapy Modalities; Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physiotherapy program (Experimental): Physiotherapy program and usual drugs
  Interventions: Behavioral: Physiotherapy
- Home exercise program (Active Comparator): Home exercise program and usual drugs
  Interventions: Other: Home exercise program

INTERVENTIONS:
Behavioral: Physiotherapy — A program of physiotherapy including manual therapy, exercise, pain education.
  Other Names: Manual Therapy, Physical Therapy
  Arms: Physiotherapy program
Other: Home exercise program — Home exercise program
  Other Names: Therapeutic exercise
  Arms: Home exercise program

SUMMARY:
This study evaluates the effectiveness of physiotherapy program in the treatment of cluster headaches. Half of participants will receive a program of physiotherapy and usual drugs, while the other will receive an exercise program and usual drugs.

DETAILED DESCRIPTION:
Previous studies have shown positive effects of physical therapy in patients with primary headache.

However, so far no study that assessed the effect of a physiotherapy program combined with regular medication in patients with cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* Cluster headache diagnosed

Exclusion Criteria:

* Other types of headaches.
* Neurostimulator implanted.
* Other chronic pain processes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Pain Scores on the Visual Analog Scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gil-Martínez, Master, Study Director — Hospital Universitario La Paz. AGClinic
Locations (1):
- AGClinic, Madrid, Madrid, Spain

REFERENCES:
- See also: AGClinic Advanced Physiotherapy — http://www.agclinic.es